CLINICAL TRIAL: NCT06042413
Title: Real-world and Innovative Multimodal Prediction and Prevention of Postoperative Mortality and Multi-morbidities
Brief Title: Prediction and Prevention of Postoperative Mortality and Morbidity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Senthil Sadhasivam, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY25110125; R01AG085115 (NIH)
Record Dates: First submitted 2023-09-06; First posted 2023-09-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Dementia; Postoperative Delirium (POD); Postoperative Neurocognitive Disorder; Major Adverse Cardiac and Cerebrovascular Events; Perioperative Complications; Postoperative Cognitive Decline
Keywords: MACCE; Cognitive decline; Perioperative brain health; Neurocognitive disorder; Postoperative delirium
MeSH Terms: conditions — Dementia; Emergence Delirium; Postoperative Cognitive Complications; Cognitive Dysfunction; Neurocognitive Disorders | interventions — Cognitive Training; Meditation

STUDY DESIGN:
Intervention Model Description: Up to 1,200 participants aged 65 years and older scheduled for elective cardiac or vascular surgery will be screened. Approximately 1,000 higher-risk participants (≥2.5% predicted risk of 30-day mortality or MACCE) who proceed to surgery will be included in Aim 1. Aim 1 is a pragmatic, non-randomized comparison in which approximately 500 participants receive CPC-guided preoperative prehabilitation and cognitive or behavioral interventions (Group A), and approximately 500 participants receive preoperative standard of care without CPC referral (Group B). Assignment is based on real-world clinical referral practices.
  Participants from Aim 1 who require intraoperative neurophysiological monitoring will be screened for Aim 2. Eligible participants (approximately 500) will be stratified by Aim 1 group and randomized 1:1 to reactive standard-of-care intraoperative management (Group C, n=250) or proactive bundled intraoperative interventions (Group D, n=250).
Masking Description: Participants are not blinded in Aim 1, however in the intraoperative intervention trial (Aim 2), participants and family members are blinded to the intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CPC Preoperative Intervention (Aim 1) (Experimental): Participants referred to the Center for Perioperative Care (CPC) by their surgical team will receive preoperative prehabilitation and proactive cognitive and behavioral interventions prior to surgery. Assignment to this group is not randomized and reflects real world clinical practice. Participants will receive standard intraoperative monitoring during surgery.
  Interventions: Other: Personalized CPC Prehabilitation; Behavioral: Cognitive Training; Behavioral: Meditation; Behavioral: Daily Exercise; Behavioral: Enhanced Social Support; Procedure: Intra-operative Standard of Care
- Preoperative Standard of Care (Aim 1) (Active Comparator): Participants who do not receive CPC referral will receive standard preoperative care prior to surgery. Assignment to this group is not randomized. Participants will receive standard intraoperative monitoring during surgery.
  Interventions: Procedure: Pre-operative Standard of Care; Procedure: Intra-operative Standard of Care
- Proactive Bundled Intraoperative Interventions (Aim 2) (Experimental): Participants in Aim 2 are drawn from Aim 1 participants who meet IONM eligibility. Participants requiring intraoperative neurophysiological monitoring will be randomized on the day of surgery to receive proactive bundled intraoperative interventions in addition to standard intraoperative monitoring.
  Interventions: Other: Proactive Bundle Interventions; Procedure: Intra-operative Standard of Care
- Reactive Intraoperative Standard of Care (Aim 2) (Active Comparator): Participants in Aim 2 are drawn from Aim 1 participants who meet IONM eligibility. Participants requiring intraoperative neurophysiological monitoring will be randomized on the day of surgery to receive reactive standard of care intraoperative management with routine SSEP and EEG monitoring.
  Interventions: Procedure: Intra-operative Standard of Care

INTERVENTIONS:
Other: Personalized CPC Prehabilitation — Patients referred for elective surgery will be scheduled for a preoperative evaluation (3 to 6 weeks prior to surgery) and will receive standardized and personalized assessment and prehabilitation according to UPMC disease specific algorithms
  Arms: CPC Preoperative Intervention (Aim 1)
Behavioral: Cognitive Training — Participants will be provided with access to the Lumosity (Lumos Labs) software for installation on a home device. They will be trained to navigate the touchscreen tablet and guided through an introductory series of brain exercise games focused on 5 main categories: memory, speed, attention, flexibility, and problem-solving. Patients will be asked to complete a cognitive exercise dosage of a minimum of 20 minutes a day for ≥5 days prior to their date of surgery. Research coordinators and volunteers from UPMC's Hospital Elder Life Program (HELP) will reach out to participants daily for a quick social check-in and to remind them to perform their training. Compliance data will be retrieved from the Lumosity app.
  Arms: CPC Preoperative Intervention (Aim 1)
Behavioral: Meditation — A single guided meditation session with instructions will be provided using a smart device. The meditation session will last for at least 10 minutes daily starting at least 1-week prior to surgery. If the subject does not own a smart device, one will be provided or meditation will be completed in-person or over the phone.
  Arms: CPC Preoperative Intervention (Aim 1)
Behavioral: Daily Exercise — Participants in the intervention group will meet with an occupational or physical therapist approximately 1-6 weeks before surgery who will discuss the potential benefits of exercise and give directions for an easy strength training exercise. Participants will then be provided with a video link for a guided exercise and encouraged to walk or perform a seated strength exercise for ≥ 5 minutes each day for at least 1 week before surgery and after surgery. Patient reported frequency, fitness app compliance and exercise duration with REDCap email or mobile link or over telephone will be collected before and after surgery. Patients will be cleared by an occupational or physical therapist to perform the upper-extremity exercises and will confirm the exercises are not contraindicated after surgery. An occupational or physical therapist will see subject again post-surgery to mitigate risk of injury.
  Arms: CPC Preoperative Intervention (Aim 1)
Behavioral: Enhanced Social Support — Research coordinators and volunteers from the Hospital Elder Life Program (HELP) will contact participants prior to surgery to discuss concerns, provide regular social support, and remind participants to complete assigned cognitive exercises. The role of family members and caregivers in supporting the participant will also be discussed, and their involvement will be encouraged when appropriate.
  Participants in the CPC preoperative intervention group may receive preoperative interventions to address depressive symptoms as part of CPC-guided prehabilitation, when clinically indicated.
  Arms: CPC Preoperative Intervention (Aim 1)
Other: Proactive Bundle Interventions — Participants randomized to the proactive bundled intervention group (Group D) will receive routine intraoperative SSEP and EEG monitoring and proactive optimization of intraoperative physiology, including maintaining mean arterial pressure ≥65 mmHg, adequate oxygenation, opioid sparing analgesia, and avoidance of deep anesthesia and benzodiazepines.
  If persistent focal changes in SSEP and EEG (i.e., changes in one hemisphere) occur, reactive measures will be implemented to increase cerebral perfusion, including ensuring hematocrit >30, maintaining anesthetic BIS >50-60, and initiating stroke management and thrombectomy if clinically indicated
  Arms: Proactive Bundled Intraoperative Interventions (Aim 2)
Procedure: Pre-operative Standard of Care — Participants will receive routine preoperative clinical care per institutional standard practice.
  Arms: Preoperative Standard of Care (Aim 1)
Procedure: Intra-operative Standard of Care — This includes routine intraoperative SSEP and EEG monitoring. Physician oversight and interpretation of real-time neuromonitoring data will be performed using a combined on-site and remote model at UPMC. In the event that changes in EEG or SSEP are considered significant by the oversight neurophysiologists, the surgical team will be immediately informed so that immediate appropriate action can be taken to reverse the change.

SUMMARY:
This study will contribute to creating a prospective and automated preoperative risk assessment algorithm for predicting 30-day mortality, major adverse cardiac and cerebrovascular events (MACCE), and postoperative neurocognitive outcomes following elective cardiac and vascular surgery in older adults. It will evaluate associations between perioperative factors and longer-term neurocognitive outcomes, including postoperative neurocognitive disorder and dementia. In addition, this study will assess scalable, multimodal preoperative and intraoperative interventions to improve perioperative outcomes.

This study will explore two main hypotheses:

1. Preoperative personalized prehabilitation with proactive cognitive and behavioral interventions will improve postoperative cognitive outcomes, morbidity, and mortality in high-risk elderly surgical patients.
2. Proactive bundled intraoperative interventions are superior to reactive standard of care in reducing postoperative cognitive outcomes, MACCE, and mortality.

Expected Outcome: Improved EHR algorithm will have higher predictive accuracy for MACCE and mortality while predicting postoperative cognitive outcomes.

DETAILED DESCRIPTION:
This study will cover the following two specific aims:

Aim 1. A pragmatic, non-randomized study to assess the effectiveness of preoperative personalized prehabilitation with proactive cognitive and behavioral interventions versus standard of care on reducing postoperative cognitive outcomes (including postoperative delirium within 30 days, postoperative cognitive decline, and dementia), MACCE, and mortality in high-risk surgical elderly patients (≥65 years). Our Electronic Health Record (EHR)-based automated machine-learning risk prediction algorithm for postoperative mortality and MACCE has been developed using >1.25 million surgical patients' data and implemented with superior performance to comparators. This EHR algorithm will identify approximately 1,000 patients at high risk for 30-day mortality and MACCE who proceed to surgery for Aim 1. Participants will receive either standard of care (n=500) or CPC-guided personalized preoperative prehabilitation with proactive cognitive or behavioral interventions (physical exercise, cognitive training, enhanced social support, and depression support) (n=500), based on real-world clinical referral practices rather than randomization. Cognitive assessments will be performed at baseline, discharge, and at 1, 3, 6, and 12 months.

Aim 2 Hypothesis: Proactive bundled intraoperative interventions are superior to standard intraoperative care in reducing postoperative cognitive outcomes, MACCE, and mortality.

Expected Outcome: The refined EHR-based risk prediction algorithm will demonstrate improved accuracy for predicting MACCE, mortality, and postoperative cognitive outcomes.

ELIGIBILITY:
Part I Inclusion Criteria:

* 65 years of age and older
* Identified as higher risk (≥2.5%) for 30-day mortality and MACCE based on the UPMC's Perioperative Model (EHR risk prediction algorithm)
* Scheduled for major cardiac surgeries including coronary artery bypass and valvular repair and/or vascular surgeries including carotid endarterectomy, aortic aneurysm repair, and major vascular surgeries
* RAI score ≥ 30
* Informed consent
* English speaking patients

Part II Inclusion Criteria:

* Enrolled in Aim 1 / Part I Preoperative Intervention Trial
* Scheduled for high-risk, cardiac or vascular surgery requiring intraoperative neurophysiological monitoring (IONM)
* Moderate and high risk for mortality based on Society of Thoracic Surgery score (score >4)

Part I Exclusion Criteria:

* Children (<18 years)
* Patients unable to provide consent
* Participants undergoing same day procedures or operations (discharged same day)
* Patients with severe preoperative medical diseases such as blindness or significant visual impairment, unresolved motor weakness, or any other perioperative events or complications that would have a bearing on the patient's ability to perform study tasks, neuropsychological tests, and proposed interventions

Part II Exclusion Criteria:

* Pregnant women
* Patients do not provide consent.
* Patients are unable to participate in cognitive and other behavioral assessment due to physical limitations
* Patients refuse any blood transfusions during surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02-03 (Estimated); Study Completion 2027-02-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative Delirium (POD) | At baseline screening, then up to 30 days post-operatively
  Postoperative delirium will be assessed using the Confusion Assessment Method (CAM). Participants will be classified as having delirium or not having delirium based on standard CAM criteria. A positive CAM indicates the presence of delirium.

SECONDARY OUTCOMES:
Depression | at pre-operative baseline screening, and then at post-operative months of 1, 3, 6, and 12.
  Patient Health Questionnaire (PHQ-9) will be used to assess depression symptoms. Scores range from 0 to 27, with higher scores indicating more severe depression. Scoring is as follows: 1 to 4 minimal, 5 to 9 mild, 10 to 14 moderate, 15 to 19 moderately severe, and 20 to 27 severe depression.
Dementia | Post-operative months 6 and 12.
  Dementia severity will be assessed using the Clinical Dementia Rating scale (CDR). Scores range from 0 (none) to 3 (severe).
Postoperative Cognitive Decline (POCD) | Post-operative months 1, 3, 6, and 12.
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA). Scores range from 0 to 30, with higher scores indicating better cognitive function. Postoperative cognitive decline will be defined as a decline in MoCA score compared with the preoperative baseline.
Postoperative Neurocognitive Disorder (PND) | Post-operative months 1 and 3.
  Postoperative neurocognitive disorder will be assessed based on changes from preoperative baseline in standardized cognitive assessments, including the Montreal Cognitive Assessment (MoCA). Declines in cognitive performance relative to baseline will be used to identify postoperative neurocognitive disorder.
30-day Major Adverse Cardiac and Cerebrovascular Events (MACCE) | Within 30 days post-surgery.
  This outcome measures whether a participant experiences any major adverse cardiac or cerebrovascular event within 30 days after surgery. Events included in this composite outcome are death from any cause, myocardial infarction (heart attack), stroke, or cardiac arrest. Participants will be counted once if they experience one or more of these events during the 30 day postoperative period.
Acute Kidney Injury (AKI) | During index hospitalization, up to 30 days post-operatively.
  Incidence of postoperative acute kidney injury based on changes in serum creatinine during the index hospitalization, consistent with standard clinical criteria.
Major Adverse Limb Events (MALE) | Post-operative months 1, 3, 6, and 12.
  Incidence of major adverse limb events including surgical or catheter-based revascularization or amputation. MALE includes any open surgical revascularization procedure (i.e., femoral endarterectomy, bypass surgery, thrombectomy or embolectomy, etc), catheter directed lysis to the lower extremities, and above ankle amputation.
Postoperative Stroke | Within 30 days post-surgery.
  Incidence of postoperative stroke confirmed by clinical diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Senthilkumar Sadhasivam, MD, MPH, MBA, Principal Investigator — University of Pittsburgh; Amy Monroe, MPH, MBA, Study Director — University of Pittsburgh
Locations (5):
- United States (5):
  - UPMC Montefiore Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Mercy Hospital, Pittsburgh, Pennsylvania
  - UPMC Passavant Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No